CLINICAL TRIAL: NCT03383497
Title: The Clinical Profile of Parkinson Disease in Egypt: A Retrospective Cohort Study
Brief Title: The Clinical Profile of Parkinson Disease in Egypt
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hatem Samir Shehata, Professor, Cairo University
Other Study IDs: CU 816
Record Dates: First submitted 2016-09-12; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Idiopathic Parkinson Disease
- Other Parkinsonian syndromes

SUMMARY:
Multi-center, retrospective observational cohort study in 4 tertiary referral centers in Cairo over the period from 2004 to 2016.

Study population. including all patients with idiopathic Parkinson disease attending. Patients were diagnosed in accordance to the United Kingdom - Parkinson Disease Society Brain Bank criteria.

DETAILED DESCRIPTION:
Retrospective, observational study that involve Medical Record Review (MRR). Data extraction and collection from medical records was organized through an electronic structured data collection form by two of authors (H.S and N.S).

The abstraction documents included; patient's age, sex, family history, age at onset, type and side of motor symptoms onset, associated non-motor manifestations. Moreover; management plan, drug history, outcome and disease progression were also verified and recorded.

During medical record reviewing (MRR); any missing documentation or poorly recorded information was managed by deleting the case.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Parkinsonian syndromes

Exclusion Criteria:

* Records with missing operationalized variables from patient records

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinsonian syndromes
Sampling Method: Non-Probability Sample
Enrollment: 1237 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
time to L-Dopa start | 6 - 12 months
  The time to L-Dopa start from symptoms onset in relation to time of Diagnosis

IPD SHARING:
Plan to Share IPD: Undecided